CLINICAL TRIAL: NCT07169539
Title: SerenApp Project: Protocol for a Pilot Study and Co-Creation of a Digital Tool for Psychological Support in Women Under Follow-Up and Breast Cancer Survivors
Brief Title: Digital Tool for Psychological Support in Women With Breast Cancer
Acronym: SerenApp
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Costa del Sol (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI24/01193
Record Dates: First submitted 2025-08-28; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Breast cancer survivors; Digital psychological intervention; eHealth; Mobile app; Co-creation; Effectiveness; Cost-effectiveness
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This pilot randomized controlled trial will assign participants in parallel to either the intervention group (access to SerenApp for 8 weeks) or the control group (usual oncological follow-up). The design allows comparison of psychological, usability, and health outcomes between groups to assess feasibility and potential effectiveness of the digital intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SerenApp Intervention (Experimental): Participants in this group will receive access to SerenApp for 8 weeks. SerenApp is a co-designed digital mental health application for breast cancer survivors, aimed at reducing stress, anxiety, and depressive symptoms, and enhancing coping strategies and empowerment. Participants will be encouraged to engage with the app modules during the study period and will complete baseline and post-intervention assessments, including validated psychological and usability measures.
  Interventions: Device: SerenApp Digital Psychological Intervention
- Usual Oncological Follow-up (No Intervention): Participants in this group will continue to receive standard oncological follow-up care according to routine clinical practice, without access to SerenApp during the study period. They will complete the same baseline and post-intervention assessments as the intervention group, which will allow comparison of psychological, quality of life, and healthcare resource outcomes.

INTERVENTIONS:
Device: SerenApp Digital Psychological Intervention — SerenApp is a co-created, personalized digital intervention designed to support the mental health of women in breast cancer follow-up or survivorship. The app includes modules targeting stress coping, anxiety, and depression, delivered via smartphone or computer. Content and functionalities were developed collaboratively with patients and healthcare professionals, ensuring usability, clinical relevance, and adherence to regulatory and ethical standards. The intervention is intended for self-guided use over eight weeks, with monitoring of engagement, completion, and user satisfaction.
  Arms: SerenApp Intervention

SUMMARY:
This study will design, test, and evaluate SerenApp, a digital health tool created to support women after completing treatment for breast cancer. Many women live for many years after breast cancer, but a large number continue to experience emotional difficulties such as anxiety, sadness, stress, or fear of the cancer coming back. These problems can strongly affect quality of life and are often not addressed during routine medical visits.

SerenApp is being developed as a safe, easy-to-use mobile application that provides psychological support and practical resources to help breast cancer survivors manage these challenges. What makes this project different is that the app will be created together with patients and healthcare professionals, to ensure that it responds to real needs and is adapted to the public health system in Spain.

The main questions of the study are:

Can SerenApp help women feel less anxious, depressed, or stressed and improve their overall quality of life?

Will women and professionals find the app useful, acceptable, and easy to use?

Could this digital tool reduce the need for additional healthcare resources and be cost-effective for the health system?

DETAILED DESCRIPTION:
The project has two main parts:

Co-creation phase:

Women who have had breast cancer and healthcare providers (such as oncologists, nurses, and psychologists) will participate in workshops and group discussions.

They will share their experiences, identify needs, and help design the functions and content of the app.

This ensures that the final product is adapted to what patients and professionals really want and need.

Pilot clinical study:

Women who have finished their breast cancer treatment will be invited to join the study.

Participants will be randomly assigned to one of two groups:

Intervention group: Women will use SerenApp for 8 weeks. The app includes exercises, information, and resources to help manage emotions, improve coping strategies, and feel more in control of their health.

Control group: Women will continue with their usual follow-up care.

All participants will complete questionnaires at the beginning and end of the study to measure emotional well-being, quality of life, satisfaction with care, and use of healthcare services.

After the 8 weeks, some women will take part in group interviews to share their opinions and experiences using the app.

By combining patient and professional input with scientific evaluation, this project will test whether SerenApp is a feasible and effective way to provide psychological support to breast cancer survivors. If it works as expected, SerenApp could become a valuable tool for women, families, and health services, offering accessible, evidence-based support to improve emotional well-being after cancer.

ELIGIBILITY:
Inclusion Criteria:

Women aged ≥18 years.

History of breast cancer with completion of primary treatment (surgery, chemotherapy, and/or radiotherapy), currently in follow-up.

Access to a smartphone or tablet with internet connection.

Ability to understand and provide written informed consent.

Sufficient knowledge of Spanish to use the app and complete questionnaires.

Exclusion Criteria:

Current recurrence or metastatic breast cancer.

Severe cognitive impairment or psychiatric disorder that may interfere with participation (e.g., psychosis, severe dementia).

Concurrent participation in another psychosocial intervention study.

Lack of access to digital devices or inability to use mobile applications.

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Stress Coping Strategies | Baseline (T0) and 8 weeks (T1)
  The CAEPO assesses cognitive and behavioral coping strategies used by oncology patients to manage stress related to their disease. It includes 40 items across seven subscales: Confrontation and Active Fighting, Self-Control and Emotional Control, Seeking Social Support, Anxiety and Anxious Worry, Passivity and Passive Resignation, Escape and Distancing, and Denial. Each item is rated on a 4-point Likert scale (0-3), with higher scores indicating greater use of each coping strategy.
Change in Anxiety Symptoms | Baseline (T0, before intervention) and 8 weeks post-intervention (T1)
  Measured using the Hospital Anxiety and Depression Scale - Anxiety subscale (HADS-A), this outcome evaluates changes in anxiety symptom severity in breast cancer survivors. The HADS-A consists of 7 items rated on a 0-3 Likert scale, with total scores ranging from 0 to 21. Higher scores indicate greater anxiety symptoms.
Change in Depressive Symptoms | Baseline (T0) and 8 weeks (T1).
  Depressive symptoms will be assessed with the Patient Health Questionnaire-9 (PHQ-9), a validated 9-item scale widely used in oncology and primary care. Higher scores indicate more severe depression.
  Total Score: 0-27

SECONDARY OUTCOMES:
Change in Health-Related Quality of Life | Baseline (T0) and 8 weeks (T1)
  Measured with the EQ-5D-5L, a standardized instrument for assessing health status across 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression Scale: Each of 5 dimensions rated from 1 (no problems) to 5 (extreme problems) Interpretation: Higher scores indicate better health-related quality of life (better outcome)
Usability of SerenApp | 8 weeks (T1, post-intervention only).
  Measured with the System Usability Scale (SUS), a validated 10-item scale assessing usability and acceptability of digital interventions. Scale: 0-100 Interpretation: Higher scores indicate better usability and acceptability (better outcome)
Satisfaction with Care | 8 weeks (T1)
  Measured with the Client Satisfaction Questionnaire-8 (CSQ-8), a validated tool assessing satisfaction with the intervention and overall care.
  Scale: 1-4 per item across 8 items Total Score: 8-32 Interpretation: Higher scores indicate greater satisfaction with care and the intervention (better outcome)

OTHER OUTCOMES:
Healthcare Resource Use and Cost-effectiveness | Baseline (T0) and 8 weeks (T1)
  Resource use will be collected with the Client Service Receipt Inventory (CSRI), complemented with economic evaluation measures, to estimate cost-effectiveness of SerenApp compared to usual follow-up.
  Scale: Not standardized; costs reported in monetary units Interpretation: Lower costs with equivalent or improved outcomes indicate better cost-effectiveness
Adherence to the Intervention | Continuously during the 8-week intervention period
  Measured with the Mobile Application Rating Scale (MARS) and app usage metrics (logins, time spent, module completion rates).
  MARS Scale: Typically 1-5 per item Usage Metrics: Number of logins, time spent, module completion rates Interpretation: Higher scores and greater engagement indicate better adherence (better outcome)
Qualitative Experiences, Barriers, and Facilitators | After 8 weeks (T1)
  Explored through post-intervention focus groups with participants and healthcare professionals, analyzed using qualitative methods to identify barriers, facilitators, and perceived benefits.
  Scale: Not applicable (qualitative analysis) Interpretation: Themes are identified through focus group discussions; no numerical scoring

CONTACTS AND LOCATIONS:
Overall Officials: Irene Zarcos-Pedrinaci, PhD, Principal Investigator — Hospital Universitario Costa del Sol
Locations (2):
- Spain (2):
  - Hospital Universitario Costa del Sol, Marbella, Malaga
  - Servicio Canario de la Salud, Santa Cruz de Tenerife

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset containing individual participant data underlying the primary and secondary outcome measures will be shared. Supporting documentation will include the study protocol and the statistical analysis plan. If feasible, analytic code will also be provided. No identifying information will be disclosed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available 12 months after publication of primary results, for a minimum of 5 years
Access Criteria: Researchers may request access by submitting a methodologically sound proposal to the study team. Approval will be required prior to data release
URL: http://www.serenapp.org